CLINICAL TRIAL: NCT01784835
Title: Early Exposure to OMT Prevents Long LOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEO-02
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Prematurity
Keywords: Osteopathic manipulative treatment; neonatology; neonatal care; prematurity; complementary and alternative medicine; length of stay
MeSH Terms: conditions — Premature Birth | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- control (Other): patients under standard medical care
  Interventions: Other: Usual care
- OMT (Experimental): patients under usual medical care plus osteopathic treatment
  Interventions: Other: osteopathic manipulative treatment

INTERVENTIONS:
Other: osteopathic manipulative treatment — Patients from this group received osteopathic treatments twice a week for the entire length of stay in the unit.
  Arms: OMT
Other: Usual care — Patients from control group received standard care plus osteopathic evaluation only, according to the same schedule as the study group.
  Arms: control

SUMMARY:
The application of osteopathic manipulative treatment (OMT) in preterm infants has been demonstrated to be effective in reducing length of stay (LOS). The scope of the present study is to investigate the association between earlier exposure to OMT and reduction of LOS in premature infants

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born at age between 29 and 37 weeks
* osteopathic treatment performed < 14 days after birth
* preterms born in the same hospital

Exclusion Criteria:

* Gestational age < 29 weeks
* Gestational age > 37 weeks
* First OMT performed after 14 days from birth
* genetic disorders
* congenital disorders
* cardiovascular abnormalities
* proven or suspected necrotized enterocolitis with or without gastrointestinal perforation proven or suspected abdominal obstruction
* pre/post surgery patients
* pneumoperitoneum
* atelectasis
* Newborn from an HIV seropositive/drug addicted mother
* respiratory disorders
* transferred to/from other hospital
* admitted for preterminal comfort care (defined as neither intubation nor cardio-respiratory resuscitation)

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of days of LOS | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

SECONDARY OUTCOMES:
effectiveness of OMT considering different lag time between birth and the first OMT | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Macerata Hospital, Macerata, Macerata, Italy

REFERENCES:
- [Background] Pizzolorusso G, Turi P, Barlafante G, Cerritelli F, Renzetti C, Cozzolino V, D'Orazio M, Fusilli P, Carinci F, D'Incecco C. Effect of osteopathic manipulative treatment on gastrointestinal function and length of stay of preterm infants: an exploratory study. Chiropr Man Therap. 2011 Jun 28;19(1):15. doi: 10.1186/2045-709X-19-15. PMID 21711535